CLINICAL TRIAL: NCT00360048
Title: Oxytocin Effects on Cytokines and Endocrine Parameters After LPS Induced Systemic Inflammatory Effects in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Other Study IDs: 2006-000246-39; EK-Nr.: 014/2006
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Sepsis
Keywords: oxytocin; tnf; sepsis; lps
MeSH Terms: conditions — Sepsis; Van der Woude syndrome | interventions — Oxytocin

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: oxytocin

SUMMARY:
The aim of this study is to determine if oxytocin administration is able to blunt LPS induced increase of cytokines (TNF-α) and if there is a change in the endocrine response after lipopolysaccharide administration in humans.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older with no disease history
* Written informed consent

Exclusion Criteria:

* Receiving any medication
* Probands who suffer from infectious disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-08

PRIMARY OUTCOMES:
TNF-alpha | six hours

SECONDARY OUTCOMES:
ACTH, cortisol, procalcitonin, IL-1ra, IL-4, IL-6, MIP-1alpha, MIP-1 beta, MCP-1, IP-10, VEGF, body temperature, BNP, Ghrelin, | six hours

CONTACTS AND LOCATIONS:
Overall Officials: Martin Clodi, MD, Associate Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Vila G, Riedl M, Resl M, van der Lely AJ, Hofland LJ, Clodi M, Luger A. Systemic administration of oxytocin reduces basal and lipopolysaccharide-induced ghrelin levels in healthy men. J Endocrinol. 2009 Oct;203(1):175-9. doi: 10.1677/JOE-09-0227. Epub 2009 Jul 8. PMID 19587265